CLINICAL TRIAL: NCT03409094
Title: A Study on Ocular Biometry Measurement of Schoolchildren and Adolescents in China
Brief Title: Dongguan Eye Study of Schoolchildren and Adolescents（DESSA）
Status: Withdrawn | Type: Observational
Why Stopped: equipments and staff are unavailable.
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiulan Zhang, Vice Director of Glaucoma Department,Director of Clinical Research Center, Director of Institution of Drug Clinical Trials, Sun Yat-sen University
Other Study IDs: 2017KYPJ119
Record Dates: First submitted 2018-01-17; First posted 2018-01-24 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Child Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a study to report the change of ocular biometry of schoolchildren and adolescents as well as its association with birth parameters in China.

ELIGIBILITY:
Inclusion Criteria:

* Schoolchildren and adolescents aged 7 to18 years in Dongguan
* Parents are willing to sign the informed written consent.

Exclusion Criteria:

* Those without informed written consent or unable to obey the study procedures

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Schoolchildren and adolescents ranging from 7 to 18 years old in Dongguan.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Changes of ocular fundus parameter in schoolchildren and adolescents | 3 years
  Record the change of retinal thickness during the follow-up periods.

SECONDARY OUTCOMES:
Changes of ocular biometry measurement in schoolchildren and adolescents | 3 years
  Record the change of choroidal thickness during the follow-up periods.
Changes of ocular anterior segment in schoolchildren and adolescents | 3 years
  Record the change of corneal thickness during the follow-up periods.

CONTACTS AND LOCATIONS:
Overall Officials: Xiulan Zhang, MD,PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No